CLINICAL TRIAL: NCT06640166
Title: Encorafenib + Cetuximab Beyond Progression in Combination With FOLFIRI in Patients With BRAF V600E Mutated Metastatic Colorectal Cancer Progressing on Encorafenib + Cetuximab.
Acronym: ECLYPse
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Pierre Fabre Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6070; 2023-508615-24-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-07; First posted 2024-10-15 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-10

CONDITIONS: Colorectal Carcinoma; Colorectal Neoplasms; Colorectal Tumor; Colorectal Adenocarcinoma; Colorectal Cancer (CRC); Colorectal Cancer; Colon Cancer; Colon Adenocarcinoma; Colon Carcinoma; Colon Neoplasm
Keywords: BRAF; V600E; encorafenib; cetuximab; colorectal cancer; FOLFIRI; BRAF V600E
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — encorafenib; Cetuximab; IFL protocol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- encorafenib+cetuximab+FOLFIRI (Experimental): Encorafenib plus cetuximab beyond progression in combination with irinotecan-based doublet chemoterapy (FOLFIRI)
  Interventions: Drug: encorafenib + cetuximab + FOLFIRI

INTERVENTIONS:
Drug: encorafenib + cetuximab + FOLFIRI — encorafenib plus cetuximab beyond progression in combination with irinotecan-based doublet chemoterapy (FOLFIRI) as follows:
  * encorafenib 300 mg (75 mgx4 hard capsules) orally once daily;
  * cetuximab 500 mg/sqm iv every 14 days;
  * FOLFIRI iv every 14 days (Irinotecan 180 mg/sqm, Folinic Acid 400 mg/sqm, 5Fluorouracil 400 mg/sqm iv bolus and 2400 mg/sqm iv continuous infusion over 46-48 hours).
  Other Names: encorafenib; cetuximab; FOLFIRI

SUMMARY:
The aim of this study is to determine the activity of encorafenib plus cetuximab in combination with FOLFIRI in patients with BRAF V600E mutated metastatic colorectal cancer progressing on encorafenib plus cetuximab administered in second line.

DETAILED DESCRIPTION:
This is a prospective, multicentre, phase II single-arm trial, evaluating encorafenib plus cetuximab beyond progression in combination with irinotecan-based doublet chemotherapy (FOLFIRI) in patients affected by BRAF V600E mutated metatstic colorectal cancer progressing on encorafenib plus cetuximab administered in second line.

Eligible patients are:

* affected by BRAF V600E mutated metastatic colorectal cancer;
* progressing on encorafenib plus cetuximab administered in second line;
* achieved complete response, or partial response, or stable disease lasting more than 3 moths, as best response to encorafenib plus cetuximab administered in second line.

All patients eligible according to inclusion and exclusion criteria will receive encorafenib plus cetuximab beyond progression in combination with irinotecan-based doublet chemoterapy (FOLFIRI) as follows:

* encorafenib 300 mg (75 mgx4 hard capsules) orally once daily;
* cetuximab 500 mg/sqm iv every 14 days;
* FOLFIRI iv every 14 days (Irinotecan 180 mg/sqm, Folinic Acid 400 mg/sqm, 5Fluorouracil 400 mg/sqm iv bolus and 2400 mg/sqm iv continuous infusion over 46-48 hours).

Treatment will be administered until disease progression, unacceptable toxic effects, withdrawal of consent, or death.

The primary end point of this trial is investigator-assessed 6-month progression free survival rate and is defined as the proportion of patients alive and progression-free by the 6-month time point from start of investigational treatment (encorafenib plus cetuximab beyond progression in combination with FOLFIRI).

ELIGIBILITY:
Inclusion Criteria:

* written informed consent to study procedures;
* age ≥ 18 years;
* histologically or cytologically confirmed diagnosis of colorectal adenocarcinoma;
* radiological evidence of metastatic disease;
* evidence of measurable disease according to RECIST 1.1 criteria;
* presence of BRAF V600E mutation in tumor tissue (primary CRC and/or related metastasis) as previously determined by a local assay at any time prior to screening (only PCR and NGS-based local assays results will be acceptable);
* disease progression while on treatment with EC received in 2nd line setting

  * EC administered after disease relapse during treatment or within 6 months following adjuvant therapy will be second line;
  * maintenance therapy given in the metastatic setting after a first line doublet or triplet chemotherapy will not be considered a separate regimen;
* best response to previous treatment with EC: CR, PR or SD lasting for at least 3 months.
* patient fit for a subsequent treatment line with FOLFIRI. Patients exposed to irinotecan and fluoropyrimidines during previous line for metastatic disease are eligible, provided that the patient has recovered from G3 toxicity;
* life expectancy ≥ 3 months;
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≤1.
* Adequate bone marrow function at screening:

  * Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L;
  * Platelets ≥ 100 × 10^9/L;
  * Hemoglobin ≥ 9.0 g/dL;
  * Note: Transfusions will be allowed to achieve this. Transfusions will be permitted provided that the patient has not received more than 2 units red blood cells in the prior 4 weeks to achieve this criteria.
* Adequate renal function at screening: serum creatinine ≤ 1.5 × upper limit of normal (ULN), or calculated by Cockroft-Gault formula, or directly measured creatinine clearance ≥ 50 mL/min at screening.
* Adequate hepatic function at screening:

  * serum total bilirubin ≤ 1.5 × ULN;
  * alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤ 2.5 × ULN, or ≤ 5 × ULN in presence of liver metastases.
* Adequate cardiac function characterized by the following at screening: QT interval corrected for heart rate using Fridericia's formula (QTcF) value ≤480 msec.
* Availability of treatment-naïve, archival FFPE tumor tissue sample.
* Ability to take oral medications.
* Male subjects with female partners of childbearing potential must be willing to use adequate contraception, starting with the first dose of study therapy through 180 days after the last dose of treatment. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
* Women of childbearing potential must have a negative blood or urine pregnancy test at the baseline visit.
* Female subjects of childbearing potential must be willing to use an adequate method of contraception, for the course of the study starting with the first dose of study therapy through 180 days after the last dose of treatment. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
* Will and ability to comply with the protocol.

Exclusion Criteria:

* patients experiencing PD as best response to EC;
* patients with specific BRAFi/AntiEGFR contraindications;
* patients with specific irinotecan or fluoropyrimidines contraindications;
* patients with DPYD deficiency;
* life expectancy ≤3 months;
* ECOG PS >1.
* Any of the following in the 6 months prior to treatment start: myocardial infarction, acute coronary syndromes (including unstable angina, coronary artery bypass graft [CABG], coronary angioplasty or stenting), congestive heart failure (≥ New York Heart Association Classification Class II), serious cardiac arrhythmia (except atrial fibrillation and appropriately controlled paroxysmal supraventricular tachycardia), cerebrovascular accident, symptomatic pulmonary embolism.
* Congenital long QT syndrome.
* Impaired gastrointestinal function or disease that may significantly alter the absorption of encorafenib (uncontrolled vomiting, malabsorption syndrome, small bowel resection with decreased intestinal absorption).
* Uncontrolled coagulopathy.
* Patients has a known history of Gilbert's syndrome or is known to have any of the following genotypes: UGT1A1*6/*6, UGT1A1*28/*28, or UGT1A1*6/*28.
* Active infection requiring systemic therapy.
* Known history of acute or chronic pancreatitis.
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive).
* Symptomatic brain metastasis or leptomeningeal disease. Prior hypersensitivity or toxicity that would suggest an inability to tolerate administration of the planned dose of investigational products.
* Residual CTCAE > Grade 2 toxicity from any prior anticancer therapy, with the exception of alopecia or neuropathy.
* Any concomitant drugs contraindicated for use with the trial drugs according to the product information of the pharmaceutical companies, including current treatment with a non-topical medication known to be a strong inhibitor of cytochrome P450 (CYP) 3A4 ≤ 1 week prior to the start of study treatment.
* Concomitant use of St. John's Wort (hypericum perforatum).
* Other severe, acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or that may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient an inappropriate candidate for the study.
* Concurrent or previous other malignancy within the past 3 years, with the exception of effectively treated squamous cell or basal cell skin cancer, melanoma in situ, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in situ of the cervix, carcinoma in situ of the colon or rectum, or other noninvasive or indolent malignancy without Sponsor approval.
* Pregnant or lactating women. Women of childbearing potential with either a positive or no pregnancy test at baseline. Postmenopausal women must have been amenorrhoeic for at least 12 months to be considered of non-childbearing potential. Sexually active males and females (of childbearing potential) unwilling to practice contraception during the study and until 180 days after the last trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
6-month Progression Free Survival rate | 6 months after the enrollment of the last patient.
  The proportion of patients alive and progression-free by the 6-month time point from start of investigational treatment (encorafenib plus cetuximab beyond progression in combination with FOLFIRI). Progression free survival is defined as the time elapsed between start of investigational treatment and the date of first event (progression or death, whichever occurs first).

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 6 months after the enrollment of the last patient.
  Time elapsed from start of investigational treatment to the documentation of investigator-assessed disease progression, according to RECIST 1.1, or death due to any cause, whichever occurs first.
Overall Survival (OS) | 6 months after the enrollment of the last patient.
  Time elapsed from start of investigational treatment to the date of death due to any cause.
Duration of response (DOR) | 6 months after the enrollment of the last patient.
  Time from response, in patients who achieve partial response (PR) or complete response (CR), to disease progression or death.
Overall Response Rate (ORR) | 6 months after the enrollment of the last patient.
  Percentage of patients who achieve PR or CR as measured by RECIST 1.1 criteria.
Disease Control Rate (DCR) | 6 months after the enrollment of the last patient.
  percentage of patients who achieve PR, CR or stable disease (SD) as measured by RECIST 1.1 criteria.
Rate of adverse events | 6 months after the enrollment of the last patient.
  Number of participants with treatment-related adverse events (graded according to NCI CTCAE version 4.03)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Alessandra Calegari, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (3):
- Italy (3):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli, IRCCS, Roma
  - Ospedale Cardinale G. Panico, Tricase

IPD SHARING:
Plan to Share IPD: No